CLINICAL TRIAL: NCT01324804
Title: Target Tissue Concentration of Standard Antibiotic Treatment in Coronary Artery Bypass Grafting Using Left Internal Mammary Artery
Brief Title: Antibiotic Concentration in Internal Mammary Graft Preparation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Medical University of Vienna, Department of Cardiothoracic- and Vascular Anaesthesia & Intensive Care Medicine
Other Study IDs: Version 1.1 - 19.11.2009
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2009-12

CONDITIONS: Coronary Heart Disease; Surgical Wound Infection
Keywords: postoperative wound healing
MeSH Terms: conditions — Coronary Disease; Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CABG - subjects: only one group

SUMMARY:
The negative effect of internal mammary harvesting on sternal perfusion is well known, especially in diabetic subjects. Microdialysis previously showed increased lactate tissue concentration after mammary artery preparation. Although high antibiotic concentration is of utmost importance in this region, no study previously measured the effect of internal mammary artery harvesting on target tissue antibiotic concentration.

Study hypothesis:

Internal mammary artery harvesting imposes an additional risk for deep sternal wound infection by impairing antibiotic tissue penetration. This effect is mediated by altered perfusion patterns and may be seen in cephalosporin and/or Teicoplanin treatment.

Study objective:

To evaluate the impact of left internal mammary artery preparation on target tissue antibiotic concentration of Cefazolin and Teicoplanin during cardiac surgery

Design:

This study is designed as an observational pharmacokinetic trial. Patients are their own controls by measuring antibiotic concentration in different subcutaneous tissues.

Study population:

Patients referred for coronary artery bypass grafting to the Department of Cardiothoracic Surgery with planned unilateral left internal mammary artery preparation and a high risk profile for deep sternal wound infections will be asked to participate in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Planned coronary artery bypass grafting with unilateral internal mammary artery bypass
* Planned used of cardiopulmonary bypass

Exclusion Criteria:

* Inability to give informed consent
* Know allergy to cephalosporins, penicillin or Teicoplanin
* Re-operation
* Additional planned valve surgery
* Dialysis
* BMI > 30
* Long standing diabetes mellitus (> 7 years)
* Ejection fraction below 20% measured with transthoracic echocardiography
* Chronic severe renal insufficiency
* Childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for coronary artery bypass grafting to the Department of Cardiothoracic Surgery with planned unilateral left internal mammary artery preparation and a high risk profile for deep sternal wound infections will be asked to participate in this trial.
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2010-11

PRIMARY OUTCOMES:
- Difference of tissue concentration of Teicoplanin between left and right pre-sternal subcutaneous tissue and between the subcutaneous tissue at the tight | 10 hours
  measurement with microdialysis
- Difference of tissue concentration of Cefazolin between left and right pre-sternal subcutaneous tissue and between the subcutaneous tissue at the tight | 10 hours
  measurement with microdialysis

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria